CLINICAL TRIAL: NCT05609097
Title: PRIME HFrEF: Novel Exercise for Older Patients With Heart Failure With Reduced Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Allen, principle investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSR220112; 1R01AG075556-01A1 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF; VO2peak
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective randomized open-label blinded endpoint (PROBE) parallel-group design. Participants will be randomized to PRIME or COMBO training for an initial four weeks (Phase 1). Following this, all participants will complete an additional eight weeks of COMBO training (Phase 2). Participants will be randomized in a 1:1 ratio by an independent statistician James Patrie (permuted block randomization with block size of 4, stratified by gender), with treatment allocation revealed after baseline exercise testing. Outcomes will be assessed at baseline, four weeks and eight weeks and 36 weeks (exploratory aim 5) by a blinded assessor (UVA SoM Exercise Core Laboratory).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRIME + COMBO (Experimental): PRIME training (Phase 1), followed by 8 weeks of progressive whole-body COMBO training.
  Interventions: Other: PRIME; Other: COMBO
- COMBO only (Other): 4 weeks of standard progressive whole-body aerobic plus resistance training (COMBO) followed by 8 weeks continued COMBO training.
  Interventions: Other: COMBO

INTERVENTIONS:
Other: PRIME — PRIME is a a 'hybrid' aerobic-resistance (cardio and weights) program designed to target all major muscle groups and address the muscle limitations responsible for reduced fitness in the elderly. This occurs by minimizing the central limitations to more traditional exercise by delivering an ideal exercise stimulus to muscles in a way in which the heart is not a limiting factor. Each exercise involves contractions of specific isolated muscle groups with a moderate load, defined as 40%-50% of their maximal voluntary capacity.
  Other Names: Exercise
  Arms: PRIME + COMBO
Other: COMBO — COMBO training includes both aerobic ("cardio") and resistance ("weightlifting") exercises. The aerobic component will be done on the stationary bicycle at 10-15 min duration at a target exercise intensity of 40-50% of VO2peak. This will feel like an intensity that is fairly light to somewhat hard, progressing gradually according to tolerance up to 20 mins. Intensity will be adjusted so that the difficulty remains in the target zone. The resistance component involves eight exercises, two sets of 10 repetitions, initially prescribed at 50-60% 1 repetition max. Subject will lift about half of their predicted maximal strength, 10 times, on 2 separate occasions with a rest between. Thereafter, the difficulty will be increased by approximately 10% when difficulty drops below the target range.
  Other Names: Exercise

SUMMARY:
This study is trying to find out whether performing a hybrid aerobic-resistance exercise training program (titled PRIME: Peripheral Remodeling via Intermittent Muscular Exercise) results in better health outcomes than the traditional exercise training program (called COMBO) that is used in individuals with heart failure with reduced ejection fraction (HFrEF). Participants will be randomized (like the flip of a coin) to either PRIME (investigational) or the traditional exercise program (standard of care).

DETAILED DESCRIPTION:
This study is a two-arm, prospective randomized clinical trial with participants randomized, in a 1:1 ratio to 4 weeks of either standard progressive whole-body aerobic plus resistance training (COMBO) or PRIME training (Phase 1), followed by 8 weeks of progressive whole-body COMBO assigned to all participants (Phase 2). The objective of this study is to determine whether PRIME exercise training can outperform traditional (COMBO) exercise training to improve outcomes in HFrEF patients. The study aims to test 92 HFrEF patients (46 randomized to PRIME and 46 to COMBO training) over a 5-year period. Data will be collected at each visit and patients will return for a 6-month follow up from the date of the final visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
* Subjects may be of either sex with age > 65 years.
* Subjects must be diagnosed with HFrEF as per established echocardiographic criteria (New York Heart Association Class II-III) with an ejection fraction <45%.
* Cardiologist approve after thorough chart review and physical examination
* Hemoglobin of at least 10.0 g/dL

Exclusion Criteria:

* Progressive worsening of exercise tolerance or dyspnea at rest or on exertion over previous 3-5 days
* Significant ischemia at low exercise intensities (<2 METS or ~50 W)
* Uncontrolled diabetes (HbA1c >10%)
* Acute systemic illness of fever
* Recent embolism (in the 6 weeks)
* Deep Vein Thrombophlebitis
* Active pericarditis or myocarditis
* Severe aortic stenosis (aortic valve area <1.0 cm2)
* Regurgitant valvular heart disease requiring surgery
* Myocardial infarction within previous 3 weeks
* New onset atrial fibrillation (in the last 4 weeks)
* Resting Heart Rate >120bpm

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
VO2peak | 12 weeks
  Change in cardiorespiratory fitness (peak oxygen consumption [V̇O2peak]) after 12 weeks of training. The primary null hypothesis will test if mean change in V̇O2peak after 12 weeks of training is the same for subjects who initially undergo 4 weeks of PRIME before undergoing 8 weeks of progressive whole-body COMBO, versus subjects who undergo the whole 12 weeks of progressive COMBO. The alternative hypothesis is that the mean change in V̇O2peak after 12 weeks of training is not the same for subjects who initially undergo 4 weeks of PRIME training before undergoing 8 weeks of progressive COMBO, versus subjects who undergo the whole 12 weeks of progressive COMBO. Secondary endpoints include blood pressure, vascular function [arterial stiffness, endothelial function (FMD)] muscle characteristics and histochemistry, blood chemistry, physical fitness testing, quality of life questionnaires, and adherence.

SECONDARY OUTCOMES:
Muscular fitness | 40- weeks
  Evaluated using 1 repetition maximal strength [1RM] measured in kg units
Physical Function | 40- weeks
  Evaluated by the Senior Fitness Test scores [SFT], measured in percentile units.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Allen, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Department of Kinesiology, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Allen JD, Vanbruggen MD, Johannsen NM, Robbins JL, Credeur DP, Pieper CF, Sloane R, Earnest CP, Church TS, Ravussin E, Kraus WE, Welsch MA. PRIME: A Novel Low-Mass, High-Repetition Approach to Improve Function in Older Adults. Med Sci Sports Exerc. 2018 May;50(5):1005-1014. doi: 10.1249/MSS.0000000000001518. PMID 29232316
- [Background] Shoemaker MJ, Curtis AB, Vangsnes E, Dickinson MG. Triangulating Clinically Meaningful Change in the Six-minute Walk Test in Individuals with Chronic Heart Failure: A Systematic Review. Cardiopulm Phys Ther J. 2012 Sep;23(3):5-15. PMID 22993497
- [Background] Allen JD, Robbins JL, Vanbruggen MD, Credeur DP, Johannsen NM, Earnest CP, Pieper CF, Johnson JL, Church TS, Ravussin E, Kraus WE, Welsch MA. Unlocking the barriers to improved functional capacity in the elderly: rationale and design for the "Fit for Life trial". Contemp Clin Trials. 2013 Sep;36(1):266-75. doi: 10.1016/j.cct.2013.07.007. Epub 2013 Jul 27. PMID 23900005
- [Background] Rickli H, Kiowski W, Brehm M, Weilenmann D, Schalcher C, Bernheim A, Oechslin E, Brunner-La Rocca HP. Combining low-intensity and maximal exercise test results improves prognostic prediction in chronic heart failure. J Am Coll Cardiol. 2003 Jul 2;42(1):116-22. doi: 10.1016/s0735-1097(03)00502-3. PMID 12849670
- [Background] Angadi SS, Jarrett CL, Sherif M, Gaesser GA, Mookadam F. The effect of exercise training on biventricular myocardial strain in heart failure with preserved ejection fraction. ESC Heart Fail. 2017 Aug;4(3):356-359. doi: 10.1002/ehf2.12149. Epub 2017 Mar 16. PMID 28772048
- [Background] Angadi SS, Mookadam F, Lee CD, Tucker WJ, Haykowsky MJ, Gaesser GA. High-intensity interval training vs. moderate-intensity continuous exercise training in heart failure with preserved ejection fraction: a pilot study. J Appl Physiol (1985). 2015 Sep 15;119(6):753-8. doi: 10.1152/japplphysiol.00518.2014. Epub 2014 Sep 4. PMID 25190739